CLINICAL TRIAL: NCT07398222
Title: Ultrasonographic Evaluation of Gastric Content in Fasting Volunteers and in Tirzepatide Users: an Observational and Cross-sectional Study
Brief Title: Gastric Content in Fasting Volunteers and in Tirzepatide Users: an Observational and Cross-sectional Study
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Guilherme Freitas Araujo, MD, Hospital Israelita Albert Einstein
Other Study IDs: 90834625.3.0000.0071
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Full Stomach Status
Keywords: gastric ultrasonography; tirzepatide; full stomach

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- fasting tirzepatide users: Individuals currently using the medication tirzepatide, who have fasted for at least 8 hours for solids and 2 hours for clear liquids without residues.
  Interventions: Other: Ultrasonographic evaluation of gastric content
- fasting volunteers.: Individuals not currently using the medication tirzepatide or any types of GLP-1 analogs, who have fasted for at least 8 hours for solids and 2 hours for clear liquids without residues.
  Interventions: Other: Ultrasonographic evaluation of gastric content

INTERVENTIONS:
Other: Ultrasonographic evaluation of gastric content — Ultrasonographic evaluation of gastric content

SUMMARY:
Introduction

Obesity and type 2 diabetes mellitus constitute a global public health problem. Medications with glucagon-like peptide-1 (GLP-1) receptor agonist activity are a modern therapeutic option for both diseases. Liraglutide, semaglutide, dulaglutide and tirzepatide are representatives of this drug class, whose mechanism of action results in delayed gastric emptying, reduced gastric motility and increased gastric volume.

Tirzepatide, however, presents a dual agonist action, combining GLP-1 agonism with glucose-dependent insulinotropic polypeptide (GIP) agonism.

The presence of gastric content during anaesthesia may lead to pulmonary aspiration and the development of chemical pneumonitis, a potentially devastating complication. However, when there is a risk factor for delayed gastric emptying, despite adequate fasting, the stomach may still present residual content, and bedside ultrasonography is an effective, non-invasive and rapid method to measure this content and stratify aspiration risk.

Our hypothesis is that most individuals using tirzepatide present a full stomach even after fasting times recommended in the literature.

DETAILED DESCRIPTION:
OBJECTIVES

1. Primary objective The primary objective is to evaluate the prevalence of a full stomach through gastric ultrasonography in volunteers who are using tirzepatide and have been fasting for at least 8 hours for solids and 2 hours for clear liquids.
2. Secondary objectives The secondary objectives are to evaluate whether the volunteers' demographic characteristics, duration of medication use, time elapsed since the last dose of tirzepatide, dose and dosing regimen, reason for medication use, and the presence of symptoms such as nausea, vomiting, and a sensation of gastric fullness may influence gastric emptying when these individuals are evaluated by ultrasonography.

2. STUDY DESIGN 2.1 Study design Observational, cross-sectional, non-interventional study. Study flowchart Below we present a schematic illustration of the study design.

3. STUDY POPULATION 3.1 Center and population Thirty volunteers will be included in the study, of whom 15 must be currently using tirzepatide and 15 must not be using the medication.

Potential volunteers may be invited in person, such as coworkers, individuals from their social circle, or even patients already referred to the Center for Interventional Medicine for other examinations/procedures.

The approach may also be carried out via WhatsApp message through the following invitation:

"You are being invited to participate in a study entitled 'Ultrasonographic evaluation of gastric content in fasting volunteers using Tirzepatide: an observational and cross-sectional study.' If you are using tirzepatide, we would like to invite you to participate in this study, which investigates gastric content in individuals with 8 hours of fasting through an abdominal ultrasonography examination. If you are interested in participating, please contact Dr. Guilherme Araújo at the phone number (11) 95638-2319." The process of obtaining the Informed Consent Form (ICF) will be conducted by the principal investigator or by a duly trained and delegated member of the research team, in person, prior to performing the ultrasonography examination. Thus, the consent process-namely, after understanding the study and voluntary confirmation of participation-must be obtained through a signed physical ICF before participation. After signing, the participant will receive a fully signed copy. A note will be made in the patient's medical record indicating the date on which the ICF was applied.

After inclusion in the study, gastric ultrasonography will be performed at Hospital Israelita Albert Einstein by an anesthesiologist experienced in gastric ultrasound. Images will be recorded in the PACS system (Picture Archiving and Communication System) and reviewed by a radiologist.

4. INCLUSION CRITERIA Adult individuals (age ≥ 18 years). Individuals currently using the medication tirzepatide. Individuals who have fasted for at least 8 hours for solids and 2 hours for clear liquids without residues.

4.1. Exclusion criteria Pregnant and postpartum individuals. Individuals with technical limitations for gastric content assessment by ultrasound (see definitions, section 5.3.3).

Presence of risk factors for gastroparesis (see definitions, section 3.2). Use of prokinetic medications that accelerate gastric emptying, such as bromopride, metoclopramide, and domperidone.

5.4 Sample size calculation Based on the literature (16), individuals in the control group presented residual gastric fluid areas ranging from 3 cm² to 7 cm², with a median area of 5.1 cm², which respectively correspond to 32.4 mL, 90.8 mL, and 63.1 mL of residual gastric fluid volume after 8 hours of fasting. Assuming an average increase of at least 20 mL of fluid in patients using semaglutide, with 95% confidence and 80% power, the required sample size for the study is 14 patients per group. To compensate for potential losses, the sample size will be increased by 10%, resulting in 15 volunteers in each group. Solid residue assessment will be descriptive, as any amount classifies the individual as having a full stomach. Furthermore, it is expected that individuals without risk factors for gastroparesis will present no solid residue after the recommended fasting period (8), making sample size calculation not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Individuals currently using tirzepatide.
* Individuals fasting for at least 8 hours for solids and 2 hours for clear liquids without residue.

Exclusion Criteria:

* Pregnant or postpartum individuals.
* Technical limitation for gastric ultrasound assessment.
* Presence of risk factors for gastroparesis.
* Use of prokinetic medications such as bromopride, metoclopramide or domperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty volunteers will be included, of whom 15 will be current users of tirzepatide and 15 will not be using the medication.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of the prevalence of a full stomach after fasting using gastric ultrasonography in volunteers using tirzepatide versus those not using the medication. | 1 day
  Comparison of the prevalence of a full stomach after fasting using gastric ultrasonography in volunteers using tirzepatide versus those not using the medication. The outcome is binary: a full stomach is defined as the presence of solids or clear liquid volume greater than 1.5 mL/kg.

SECONDARY OUTCOMES:
demographic characteristics | 1 day
  * Demographic characteristics
  * Dose and dosing regimen
  * Indication for medication use
  * Presence of symptoms (nausea, vomiting, gastric fullness, early satiety, abdominal pain)
  * Use of other medications

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme F Araujo, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-02-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT07398222/Prot_SAP_000.pdf